CLINICAL TRIAL: NCT01681836
Title: An Open-Label Study of Oral Nitrite and Nitrate in Healthy Normal Volunteer Adults
Brief Title: Oral Nitrite and Nitrate in Healthy Normal Volunteer Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gladwin, Mark, MD (Individual)
Responsible Party: Principal Investigator, Kara Hughan, Instructor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRO11120134
Record Dates: First submitted 2012-07-03; First posted 2012-09-10 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Focus of Study of Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral 15N-labeled sodium nitrate (Experimental): Oral sodium nitrate 1,000 mg once first, then washout followed by oral sodium nitrite 20 mg once
  Interventions: Drug: 15Nitrogen(15N)-labeled sodium nitrite; Drug: 15Nitrogen(15N)-labeled sodium nitrate
- Oral 15N-labeled sodium nitrite (Experimental): Oral sodium nitrite 20 mg once first, then washout followed by oral sodium nitrate 1,000 mg once
  Interventions: Drug: 15Nitrogen(15N)-labeled sodium nitrite; Drug: 15Nitrogen(15N)-labeled sodium nitrate

INTERVENTIONS:
Drug: 15Nitrogen(15N)-labeled sodium nitrite — 15Nitrogen(15N)-labeled sodium nitrite 20 mg once
Drug: 15Nitrogen(15N)-labeled sodium nitrate — 15Nitrogen(15N)-labeled sodium nitrate 1,000 mg once

SUMMARY:
This proposal hypothesizes that oral supplementation with sodium nitrite or nitrate will result in in vivo conversion of nitrate to nitrite and nitrite to nitric oxide with limited toxicity in the doses proposed in healthy adult normal volunteers. We utilize a powerful in vivo technique (pharmacokinetic testing) and are the first to design inorganic nitrate and nitrite capsules for cardiovascular disease.

DETAILED DESCRIPTION:
Preclinical and clinical research over the last decade has revealed the important vasoprotective effects of nitrates and nitrites with regards to reduction in blood pressure, vascular inflammation and endothelial dysfunction. New findings suggest an effect of nitrate and nitrite therapy in the regulation of glucose-insulin homeostasis. Development of an oral formulation of nitrate and nitrite salts is attractive, whereby nitrite would ensure rapid acting effects upon absorption, while the nitrate would continuously provide a slow formation of nitrite over a prolonged period of time via the enterosalivary circulation pathway.

For this reason, development of an oral formulation of nitrate and nitrite salts is attractive, whereby nitrite would ensure rapid acting effects upon absorption, while the nitrate would continuously provide a slow formation of nitrite over a prolonged period of time via the enterosalivary circulation pathway. This study aims to establish the pharmacokinetics, metabolism and interconversion of nitrate to nitrite and nitrite to nitric oxide in vivo in healthy adult normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Systolic blood pressure ≤130 and diastolic blood pressure ≤85 mm Hg

Exclusion Criteria:

* Positive urine pregnancy test or breastfeeding
* Concurrent use of medications affecting glucose or lipid metabolism
* Recent addition or change in dosing of hormonal contraceptive medications (oral contraceptive pill, intrauterine device, DepoProvera)
* Current use of ≥2 anti-hypertensive agents regardless of blood pressure control or normotensive on a single agent
* Current use of phosphodiesterase 5 inhibitors or organic nitrates
* Not stable on treatments for the prior three months or not planning to remain on current dose of medications for blood pressure, contraception, etc
* Known chronic psychiatric or medical conditions including diabetes, liver or kidney disease or obesity syndromes
* Smoker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara S Hughan, MD, Principal Investigator — University of Pittsburgh; Mark T Gladwin, MD, Study Director — University of Pittsburgh; Bret Goodpaster, PhD, Study Director — University of Pittsburgh
Locations (1):
- Montefiore Hospital of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Hughan KS, Wendell SG, Delmastro-Greenwood M, Helbling N, Corey C, Bellavia L, Potti G, Grimes G, Goodpaster B, Kim-Shapiro DB, Shiva S, Freeman BA, Gladwin MT. Conjugated Linoleic Acid Modulates Clinical Responses to Oral Nitrite and Nitrate. Hypertension. 2017 Sep;70(3):634-644. doi: 10.1161/HYPERTENSIONAHA.117.09016. PMID 28739973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult participants were recruited between October 2012 and October 2013.
Pre-assignment Details: 11 participants recruited; 11 screened; 0 excluded
Groups:
- Oral 15N-labeled Sodium Nitrate, Then Sodium Nitrite: Oral 15N-labeled sodium nitrate 1,000 mg once in first intervention period and oral 15N-labeled sodium nitrite 20 mg once in second intervention period (after washout period)
- Oral 15N-labeled Sodium Nitrite, Then Sodium Nitrate: Oral 15N-labeled sodium nitrite 20 mg once in first intervention period and oral 15N-labeled sodium nitrate 1,000 mg once in second intervention period (after washout period)
Period: First Intervention
Arm/Group | Oral 15N-labeled Sodium Nitrate, Then Sodium Nitrite | Oral 15N-labeled Sodium Nitrite, Then Sodium Nitrate
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout Period of 3-7 Days
Arm/Group | Oral 15N-labeled Sodium Nitrate, Then Sodium Nitrite | Oral 15N-labeled Sodium Nitrite, Then Sodium Nitrate
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Oral 15N-labeled Sodium Nitrate, Then Sodium Nitrite | Oral 15N-labeled Sodium Nitrite, Then Sodium Nitrate
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to received oral 15N-labeled sodium nitrate first and sodium nitrite first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 30.4 [21 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 122 (9.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 75 (9.3)
Mean arterial pressure [Mean (Standard Deviation); unit: mmHg] | 91 (6.8)
Methemoglobin [Mean (Standard Deviation); unit: percentage level of methemoglobin] | 1.0 (0.2)

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Nitrate Concentration Over 24 Hour Study Period
Description: "Post-doses" refers to that subjects will receive a single dose of each study drug, oral 15Nitrogen(15N)-labeled sodium nitrate and nitrite, in random order, separated by a 3-7 day washout period
Time Frame: measured at 0 (baseline), 0.5, 1, 2, 3, 6 and 24 hours post-doses
Measure: Mean (Standard Error); unit: microMolar (microM)
Groups:
- Oral 15N-labeled Sodium Nitrate: Oral 15N-labeled sodium nitrate 1,000 mg once in either first intervention period or second intervention period
- Oral 15N-labeled Sodium Nitrite: Oral 15N-labeled sodium nitrite 20 mg once in either first intervention period or second intervention period
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
microMolar (microM) | 769 (38) | 41 (3.7)

2. Primary Outcome: Peak Plasma Nitrite Concentration Over 24 Hour Study Period
Description: as for outcome 1
Time Frame: measured at 0 (baseline), 0.5, 1, 2, 3, 6 and 24 hours post-doses
Measure: Mean (Standard Error); unit: microM
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
microM | 0.51 (0.1) | 5.5 (0.7)

3. Primary Outcome: Peak Red Blood Cell (RBC) Iron-nitrosyl Hemoglobin (NO-Hb) Concentrations Over 24 Hour Study Period
Description: as for outcome 1
Time Frame: measured at 0 (baseline), 0.5, 1, 2, 3, 6 and 24 hours post-doses
Measure: Mean (Standard Error); unit: microMolar
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
microMolar | NA (NA) — not detectable | 1.04 (0.22)

4. Secondary Outcome: Peak Percentage Level of Methemoglobin Over 24 Hour Study Period
Description: "Post-doses" refers to that subjects will receive a single dose of each study drug, oral 15N-labeled sodium nitrate and nitrite, in random order, separated by a 3-7 day washout period
Time Frame: measured at 0 (baseline), 0.5, 1, 2, 3, 6 and 24 hours post-doses
Measure: Mean (Standard Error); unit: percentage level
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
percentage level | 1.24 (0.08) | 1.59 (0.09)

5. Secondary Outcome: Peak Change in Mean Arterial Pressure Over 24 Hour Study Period
Description: "Post-dose" refers to that subjects will receive a single dose of each study drug, oral 15N-labeled sodium nitrate and nitrite, in random order, separated by a 3-7 day washout period
Time Frame: measured at 0 (baseline) then every 15 minutes during the first 2 hours post-dose, then at 3, 6, and 24 hours post-dose, change at 0.75 hours reported
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
mmHg | -2.9 (2.1) | -10.4 (3.8)

6. Secondary Outcome: Peak Change in Systolic Blood Pressure Over 24 Hour Study Period
Description: as for outcome 5
Time Frame: measured at 0 (baseline) then every 15 minutes during the first 2 hours post-dose, then at 3, 6, and 24 hours post-dose, change at 1.5 hours reported
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
mmHg | -0.8 (2.9) | -12.1 (10.5)

7. Secondary Outcome: Peak Change in Diastolic Blood Pressure Over 24 Hour Study Period
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
mmHg | -6.3 (1.2) | -8.1 (6.4)

8. Secondary Outcome: Peak 15Nitrogen Nitro-conjugated Linoleic Acid (cLA) Concentrations Over 24 Hour Study Period
Description: as for outcome 5
Time Frame: measured at time 0 (trough), every 15 minutes during the first 2 hours post-dose, then at 3, 6, and 24 hours post-dose
Population: maximal at 24 hours with nitrate treatment, not detectable with nitrite treatment
Measure: Median (Full Range); unit: nanoMolar
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
nanoMolar | 0.14 [0 to 25.3] | NA [NA to NA] — not detectable

9. Secondary Outcome: Percent Platelet Activation at 6 Hours
Description: at timepoint with greatest change from 0 (trough); "Post-dose" refers to that subjects will receive a single dose of each study drug, oral 15N-labeled sodium nitrate and nitrite, in random order, separated by a 3-7 day washout period; percentage of platelets that express 2 specific markers identifying activated platelets (CD41 and CD62-P) were quantified using flow cytometry
Time Frame: measured at 0 (baseline), 6 and 24 hours post-dose
Measure: Mean (Standard Error); unit: % of platelets that are activated
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
% of platelets that are activated | 9.0 (1.7) | 8.3 (1.9)

10. Secondary Outcome: Peak Change in Heart Rate Over 24 Hour Study Period
Description: as for outcome 5
Time Frame: measured at 0 (baseline), every 15 minutes during the first 2 hours post-dose, then at 3, 6, and 24 hours post-dose, change at 1.5 hours for nitrate and 24 hours for nitrite
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Number analyzed (Participants) | 10 | 10
beats per minute | -6 (4.1) | 9 (4.4)

ADVERSE EVENTS:
Time Frame: 3-7 days after single dose of each drug
Arm/Group | Oral 15N-labeled Sodium Nitrate | Oral 15N-labeled Sodium Nitrite
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 9/10 | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral 15N-labeled Sodium Nitrate (N=10) | Oral 15N-labeled Sodium Nitrite (N=11)
Headache (Nervous system disorders) | 6 (6) | 7 (7)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dizziness (General disorders) | 0 (0) | 2 (2)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mean arterial pressure decrease >20% (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No